CLINICAL TRIAL: NCT04630457
Title: Safety and Effectiveness of Electronically Controlled Prosthetic Ankle in Patients With Transtibial Amputation
Brief Title: Safety and Effectiveness of Electronically Controlled Prosthetic Ankle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Veterans Health Service Medical Center, Seoul, Korea (Other)
Collaborators: Asan Medical Center (Other); Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Jun Yup Kim, MD, Primary Researcher, Veterans Health Service Medical Center, Seoul, Korea
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-08-011
Record Dates: First submitted 2020-09-27; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Amputation

STUDY DESIGN:
Intervention Model Description: This study is a Prospective Randomized crossover study. After randomization, the study is conducted by dividing group A (order of existing prosthesis-Meridium prosthesis-RoFT prosthesis) and B (order of existing prosthesis-RoFT prosthesis-Meridium prosthesis).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meridium-RoFT (Active Comparator): order of existing prosthesis-Meridium prosthesis-RoFT prosthesis
  Interventions: Device: Conventional ankle prosthesis; Device: Meridium® (Microprocessor ankle prosthesis); Device: RoFT® (Microprocessor ankle prosthesis)
- RoFT-Meridium (Active Comparator): order of existing prosthesis-RoFT prosthesis-Meridium prosthesis
  Interventions: Device: Conventional ankle prosthesis; Device: Meridium® (Microprocessor ankle prosthesis); Device: RoFT® (Microprocessor ankle prosthesis)

INTERVENTIONS:
Device: Conventional ankle prosthesis — At the first visit, 3D motion analysis, dynamic EMG analysis, energy consumption analysis, 6 minute walk test, Berg balance scale, Locomotor Capabilities Index, and Korean-Prosthesis Evaluation Questionnaire will be evaluated using the conventional prosthesis that the patient had.
Device: Meridium® (Microprocessor ankle prosthesis) — There are two weeks apart between each visit. Depending on the group to which the patient belongs, at the second or third visit, 3D motion analysis, dynamic EMG analysis, energy consumption analysis, 6 minute walk test, Berg balance scale, Locomotor Capabilities Index, and Korean-Prosthesis Evaluation Questionnaire will be evaluated using Meridium®. For example, if visit 2 was evaluated using Meridium®, visit 3 was evaluated using RoFT®. In another example, visit 2 is evaluated using RoFT®, while Visit 3 is evaluated using Meridium®.
Device: RoFT® (Microprocessor ankle prosthesis) — There are two weeks apart between each visit. Depending on the group to which the patient belongs, at the second or third visit, 3D motion analysis, dynamic EMG analysis, energy consumption analysis, 6 minute walk test, Berg balance scale, Locomotor Capabilities Index, and Korean-Prosthesis Evaluation Questionnaire will be evaluated using RoFT®. For example, if visit 2 was evaluated using RoFT®, visit 3 was evaluated using Meridium®. In another example, visit 2 is evaluated using Meridium®, while Visit 3 is evaluated using RoFT®.

SUMMARY:
In this study, we aim to compare the three types of prosthetic limbs: the passive prosthetic limb that the patients have been using so far, the 'RoFT', a prosthetic limb developed by the Korea Institute of Machinery & Materials, and the Meridium of Ottobock in terms of safety and effectiveness.

DETAILED DESCRIPTION:
In this study, the investigators will compare the safety and effectiveness of RoFT, a robotic ankle prosthesis developed by a Korea Institute of Machinery & Materials, Meridium of Ottobock Co., a representative commercial ankle-type robotic prosthesis, passive prosthetic limb that the patients have been using so far.

In order to compare the above three types of prostheses in terms of their effectiveness and safety, the robotic prosthesis will be evaluated after 30 minutes of familiarization after applying, and the evaluation interval using the two types of robotic prostheses will be 2 weeks to eliminate the carryover effect. For evaluation, 3D motion analysis, dynamic EMG analysis, energy consumption analysis, 6 minute walk test, Berg balance scale, Locomotor Capabilities Index, and Korean-Prosthesis Evaluation Questionnaire will be used.

For safety analysis, any kinds of safety issues including skin abrasion, bone fracture, or tendon/ligament injury due to fall down injury will be recorded and categorized for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Among patients who visited each hospital's rehabilitation department after IRB approval
2. Adults over 19 years old
3. One side transtibial amputee
4. 6 months or more from the date of amputation of the lower extremities
5. Use of the same conventional passive prosthesis for at least the last 3 months
6. Factors of K level 2 or higher (have the ability to cross low-level environmental barriers such as curbs, stairs or uneven surfaces)
7. Those who understand and agree to the test description
8. Those who did not have skin lesions on the amputation at the time of study registration
9. At least 25cm of free space from the bottom connection of the socket to the floor

Exclusion Criteria:

1. When cognitive function is deteriorated and it is impossible to independently decide to participate in research or participate in evaluation
2. Contraindications to weight-bearing of the lower extremities such as severe lower extremity joint contracture, osteoporosis, and untreated fractures
3. Patients who underwent orthopedic surgery on the lower extremities within 6 months of starting the study
4. Cardiovascular disease, venous thrombosis or heart failure, respiratory disease that may affect heart function during exercise load
5. In the presence of pain in the musculoskeletal system other than amputation that affects gait
6. Stump length over 25cm
7. Subjects judged by other testers to be unsuitable for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of Changes in Three-dimensional motion during walking | (1st visit, day 1)existing conventional prosthesis - (2nd visit, day 15)1st Microprocessor ankle prosthesis - (3rd visit, day 29) 2nd Microprocessor ankle prosthesis
  Three-dimensional motion analysis Using 8 infrared cameras and 3 force plates, set the spatial coordinates of each camera To do this, a non-linear trasformation (NLT) method is used.
  Attach 19 reflective markers for static measurement and 15 reflective markers for dynamic measurement in the standstill state on the joints and segment surfaces of the lower extremities.
  Static, Dynamic common
  * Bilateral: ■ Anterior superior iliac spine ■ On the anterior thigh ■ Lateral epicondyle of femur ■ on the lower leg ■ Lateral malleolus aligned with bimalleolar axis ■ Bisection of the proximal aspect of the posterior calcaneum ■ Dorsal surface of the left (and right) distal forefoot at the midpoint-the 2nd metatarsal head
  * Unilateral: ■ Sacrum: Mid-point on line between the PSISs
  Static only
  -Bilateral: ■ Medial epicondyle of femur ■ Medial malleolus aligned with bimalleolar axis
Analysis of Changes in dynamic EMG during walking | (1st visit, day 1)existing conventional prosthesis - (2nd visit, day 15)1st Microprocessor ankle prosthesis - (3rd visit, day 29) 2nd Microprocessor ankle prosthesis
  Dynamic EMG is calculated by measuring EMG signals by attaching surface EMG to the skin using a tape on Vastus Medialis, Rectus Femoris, Tensor Fascia Latae, Medial Hamstring, and Gluteus Maximus of both lower extremities, measuring the EMG signal, and converting it to Root mean square (RMS).
  The measured EMG signal is used to calculate the activation period and timing according to the gait cycle for each muscle, and analyze the degree of activation.
  1. Attach surface EMG to the above-mentioned muscles
  2. Muscle activation start and end points within the walking cycle
  3. Muscle activation period and RMS intergral and peak value
  4. A value obtained by dividing the RMS (Root mean square) value into 16 sections by time
  5. Comparison between healthy side and affected side
Analysis of Changes in Energy consumption during walking | (1st visit, day 1)existing conventional prosthesis - (2nd visit, day 15)1st Microprocessor ankle prosthesis - (3rd visit, day 29) 2nd Microprocessor ankle prosthesis
  * Using QUARK CPET (COSMED, Italy)
  * Perform calibration of the gas respiration analyzer 30 minutes before the start of the experiment and maintain the temperature and humidity inside the laboratory.
    * Before measurement, each amputated patient sits on a chair on the treadmill, rests for 5 minutes, and then walks on the treadmill at a comfortable pace for 3 minutes.
    * Afterwards, all amputated patients are asked to walk on the treadmill at a self-selected walking velocity.
    * The preferred speed is set to a level in which conversation is possible by deep breathing through a rating of perceived exertion (RPE).
    * Measurement is made at a preferred speed and 12% slope for 10 minutes, and walk for at least 6 minutes. If it is difficult to measure at a slope of 12% due to the subject's physiological characteristics, measure at a slope of 0%.
    * The value of rate(ml/min/kg) is obtained by averaging the value during the steady state for the last minute of the measurement section.
Analysis of Changes in 6 minute walk test | (1st visit, day 1)existing conventional prosthesis - (2nd visit, day 15)1st Microprocessor ankle prosthesis - (3rd visit, day 29) 2nd Microprocessor ankle prosthesis
  * A sub-maximal exercise test used to evaluate a patient's aerobic capacity and endurance.
  * Measure the endurance of walking by marking the distance at 30m intervals and measuring the number of round trips for 6 minutes.
Analysis of Changes in Berg balance scale(BBS) scores | (1st visit, day 1)existing conventional prosthesis - (2nd visit, day 15)1st Microprocessor ankle prosthesis - (3rd visit, day 29) 2nd Microprocessor ankle prosthesis
  * A balanced evaluation tool consisting of 14 items and a perfect score of 56
  * Item
    1. Standing while sitting
    2. Standing without help
    3. Sit by yourself without leaning
    4. Sitting while standing
    5. Moving
    6. Standing with your eyes closed
    7. Standing with both feet together
    8. Stretching and stretching arms in a standing position
    9. Lifting objects off the floor while standing
    10. Standing and looking back over both shoulders
    11. Turning 360 degrees
    12. Alternately placing both feet on the footrest while standing
    13. Standing without support with one foot in front of the other
    14. Standing on one leg
Analysis of Changes in Locomotor Capabilities Index (LCI) scores | (1st visit, day 1)existing conventional prosthesis - (2nd visit, day 15)1st Microprocessor ankle prosthesis - (3rd visit, day 29) 2nd Microprocessor ankle prosthesis
  * A scale consisting of 14 items and 56 points for the ability of patients with lower body amputation to perform activities with their will
  * Item
    ◆ Basic activity score
  * 1. Get up from the chair
  * 2. Walking in the house
  * 3. Walking on a flat surface outdoors
  * 4. Climbing stairs by holding a railing
  * 5. Go down the stairs by holding the railing
  * 6. Climb on the sidewalk block
  * 7. Going down the sidewalk block
    ◆ Advanced activity score
  * 1. Lifting objects off the floor (while standing with prosthetic feet)
  * 2. Get up from the floor (eg, if you fall)
  * 3. Walking outdoors on uneven ground (eg meadows, gravel, slopes)
  * 4. Walking outdoors in inclement weather (eg snow, rain, ice)
  * 5. Climb a few steps up the stairs without holding the railing
  * 6. Walking down the stairs a few steps without holding the railing
  * 7. Walking with objects
Analysis of Changes in Korean-Prosthesis Evaluation Questionnaire (K-PEQ) scores | (1st visit, day 1)existing conventional prosthesis - (2nd visit, day 15)1st Microprocessor ankle prosthesis - (3rd visit, day 29) 2nd Microprocessor ankle prosthesis
  * PEQ is the quality of life in various areas such as function, overall satisfaction, pain, psychosocial experience, gait and mobility, satisfaction in special situations, ability to perform daily life, will function and quality in relation to the use of the will of the amputationally disabled person. Develop to evaluate
  * PEQ is an evaluation tool conducted after 4 weeks of prosthesis and consists of a total of 86 questions in 8 areas.
  * PEQ has proven high reliability, internal consistency, content validity, and criterion validity, so it is mainly used in studies related to the will of amputation disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Yang, MD, Principal Investigator — Veterans Health Service Medical Center, Seoul, Korea
Locations (1):
- Veterans Health Service Medical Center, Seoul, Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
No IPD sharing is planned for protection of privacy.

REFERENCES:
- [Result] Han TR, Paik NJ, Im MS. Quantification of the path of center of pressure (COP) using an F-scan in-shoe transducer. Gait Posture. 1999 Dec;10(3):248-54. doi: 10.1016/s0966-6362(99)00040-5. PMID 10567757
- [Result] Patterson KK, Gage WH, Brooks D, Black SE, McIlroy WE. Evaluation of gait symmetry after stroke: a comparison of current methods and recommendations for standardization. Gait Posture. 2010 Feb;31(2):241-6. doi: 10.1016/j.gaitpost.2009.10.014. Epub 2009 Nov 22. PMID 19932621
- [Result] Collen FM, Wade DT, Bradshaw CM. Mobility after stroke: reliability of measures of impairment and disability. Int Disabil Stud. 1990 Jan-Mar;12(1):6-9. doi: 10.3109/03790799009166594. PMID 2211468
- [Result] Flansbjer UB, Holmback AM, Downham D, Patten C, Lexell J. Reliability of gait performance tests in men and women with hemiparesis after stroke. J Rehabil Med. 2005 Mar;37(2):75-82. doi: 10.1080/16501970410017215. PMID 15788341
- [Result] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Result] Bischoff HA, Stahelin HB, Monsch AU, Iversen MD, Weyh A, von Dechend M, Akos R, Conzelmann M, Dick W, Theiler R. Identifying a cut-off point for normal mobility: a comparison of the timed 'up and go' test in community-dwelling and institutionalised elderly women. Age Ageing. 2003 May;32(3):315-20. doi: 10.1093/ageing/32.3.315. PMID 12720619
- [Result] Hofheinz M, Mibs M. The Prognostic Validity of the Timed Up and Go Test With a Dual Task for Predicting the Risk of Falls in the Elderly. Gerontol Geriatr Med. 2016 Mar 16;2:2333721416637798. doi: 10.1177/2333721416637798. eCollection 2016 Jan-Dec. PMID 28138492
- [Result] Nordin E, Lindelof N, Rosendahl E, Jensen J, Lundin-Olsson L. Prognostic validity of the Timed Up-and-Go test, a modified Get-Up-and-Go test, staff's global judgement and fall history in evaluating fall risk in residential care facilities. Age Ageing. 2008 Jul;37(4):442-8. doi: 10.1093/ageing/afn101. Epub 2008 May 30. PMID 18515291
- [Result] Schmalz T, Blumentritt S, Jarasch R. Energy expenditure and biomechanical characteristics of lower limb amputee gait: the influence of prosthetic alignment and different prosthetic components. Gait Posture. 2002 Dec;16(3):255-63. doi: 10.1016/s0966-6362(02)00008-5. PMID 12443950
- [Result] Schache AG, Baker R, Vaughan CL. Differences in lower limb transverse plane joint moments during gait when expressed in two alternative reference frames. J Biomech. 2007;40(1):9-19. doi: 10.1016/j.jbiomech.2005.12.003. Epub 2006 Jan 26. PMID 16442547
- [Result] Gailey RS, Nash MS, Atchley TA, Zilmer RM, Moline-Little GR, Morris-Cresswell N, Siebert LI. The effects of prosthesis mass on metabolic cost of ambulation in non-vascular trans-tibial amputees. Prosthet Orthot Int. 1997 Apr;21(1):9-16. doi: 10.3109/03093649709164525. PMID 9141121
- [Result] Winter DA, Sidwall HG, Hobson DA. Measurement and reduction of noise in kinematics of locomotion. J Biomech. 1974 Mar;7(2):157-9. doi: 10.1016/0021-9290(74)90056-6. No abstract available. PMID 4837552